CLINICAL TRIAL: NCT02270853
Title: Incidence of Sleep Apnea Syndrome (SAS) in Patients With Bronchial Carcinoma
Brief Title: SAS in Patients With Bronchial Carcinoma
Acronym: SAS CA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 13-136
Record Dates: First submitted 2014-10-14; First posted 2014-10-21 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2016-02

CONDITIONS: Sleep Apnea Syndrome; Bronchial Carcinoma
Keywords: ApneaLink; bronchial carcinoma; sleep apnea screening
MeSH Terms: conditions — Sleep Apnea Syndromes; Carcinoma, Bronchogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- sleep apnea screening with ApneaLinkTM (Other): This is the only group in the present study. Patients with bronchial carcinoma (or reasonable suspicion) perform sleep screening with ApneaLinkTM at home or during the hospitalization.
  Interventions: Device: sleep apnea screening with ApneaLinkTM

INTERVENTIONS:
Device: sleep apnea screening with ApneaLinkTM — ApneaLink is sleep-screening tool that objectively identifies patients with sleep apnea

SUMMARY:
In this study it will be analyzed how often the sleep apnea syndrome can be observed in patients with newly diagnosed lung cancer with the help of ApneaLink device by ResMed.

DETAILED DESCRIPTION:
Determination of the SAS- frequence in patients with bronchial carcinoma. The patients will be screened at home for 1 night with the ApneaLink device by ResMed. The apneaLink device is a standard screening tool for sleep apnea in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients with reasonable suspicion of bronchial carcinoma or histologically proven bronchial carcinoma, which has not been medicated until the study entry and
* Patients with sleep apnea who had recently been diagnosed with bronchial carcinoma.

Exclusion Criteria:

* Pregnancy
* other already known malignancies or tumors
* Patients with non-invasive artificial respiration due to a chronic respiratory insufficiencies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-04; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
percent of sleep apnea in patients with bronchial carcinoma | two days
  The percent of sleep apnea in a cohort of patients with bronchial carcinoma will be evaluated. The duration of the study participation is two days.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dreher, Univ.-Prof., Principal Investigator — RWTH Aachen University Hospital
Locations (3):
- Germany (3):
  - Medizinische Klinik I Uniklinik RWTH Aachen, Aachen, North Rhine-Westphalia
  - Krankenhaus Merheim, Cologne, North Rhine-Westphalia
  - Florence-Nightingale Hospital, Düsseldorf

REFERENCES:
- [Derived] Dreher M, Kruger S, Schulze-Olden S, Keszei A, Storre JH, Woehrle H, Arzt M, Muller T. Sleep-disordered breathing in patients with newly diagnosed lung cancer. BMC Pulm Med. 2018 May 16;18(1):72. doi: 10.1186/s12890-018-0645-1. PMID 29769049